CLINICAL TRIAL: NCT05668286
Title: Comparison of the Short-term Clinical Effects of Anterior Extra-articular and Posterior Intra-articular Administration of Ultrasound-guided Steroid Injection in the Treatment of Adhesive Capsulitis. A Prospective, Randomized and Single-blind Study
Brief Title: Comparison of the Short-term Clinical Effects of Anterior Extra-articular and Posterior Intra-articular Administration of Ultrasound-guided Steroid Injection in the Treatment of Adhesive Capsulitis.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kartal City Hospital (Other)
Responsible Party: Principal Investigator, Omer Faruk Sevim, MD, Principal Investigator, Kartal City Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KartalCity-ERGUN-001
Record Dates: First submitted 2022-05-16; First posted 2022-12-29 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Adhesive Capsulitis of the Shoulder
Keywords: adhesive capsulitis; steroid injection; ultrasound-guided
MeSH Terms: conditions — Bursitis | interventions — Triamcinolone Acetonide; Prilocaine

STUDY DESIGN:
Intervention Model Description: Patients who are diagnosed with adhesive capsulitis in the orthopedic outpatient clinic will be included. Included patients will be randomly divided into two groups according to age, sex, concomitant diabetes mellitus (DM) disease and clinical stage of the disease. For randomization, stratified randomization will be applied according to the information obtained from the outpatient clinic. While patients in group 1 received an anterior extra-articular steroid injection under USG guidance, patients in group 2 received posterior intra-articular steroid injection under USG guidance.1 mL of triamcinolone acetonide and 1 mL of prilocaine hydrochloride (2%) will be injected to all patients. Patients will be first evaluated before injection, than randomized to groups and prospectively followed up by an orthopaedic surgeon who will be blinded to the groups. Evaluation will be done for pain VAS, functional status ;ASES and Quick DASH at 1,3 and 6 weeks after the injection.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- posterior intra-articular steroid injection under USG guidance (Active Comparator): Intra-articular steroid injection will be performed to the glenohumeral joint from the posterior, 2cm inferior and 2cm medial of the acromion posterolateral corner, under the guidance of USG.
  Interventions: Drug: A combination of 1 mL of triamcinolone acetonide (40 mg/mL) and 1 mL of prilocaine hydrochloride (2%)
- anterior extra-articular steroid injection under USG guidance (Active Comparator): Steroid injection will be performed from the anterior, immediately lateral to the coracoid process, to the CHL localization, to the extra-articular area under the guidance of USG.
  Interventions: Drug: A combination of 1 mL of triamcinolone acetonide (40 mg/mL) and 1 mL of prilocaine hydrochloride (2%)

INTERVENTIONS:
Drug: A combination of 1 mL of triamcinolone acetonide (40 mg/mL) and 1 mL of prilocaine hydrochloride (2%) — patients in group 1 received an anterior extra-articular steroid injection under USG guidance, patients in group 2 received posterior intra-articular steroid injection under USG guidance. A combination of 1 mL of triamcinolone acetonide (40 mg/mL) and 1 mL of prilocaine hydrochloride (2%) were injected to all patients.

SUMMARY:
In the treatment of adhesive capsulitis, conservative treatment usually gives successful results, and steroid injection is an effective method that is frequently preferred among conservative treatment modalities. However, many controversial issues have not yet been clarified in the literature, such as the location of the injection, whether into the glenohumeral joint or around the coracohumeral ligament where the most radiological findings are detected.

DETAILED DESCRIPTION:
Purpose:

To compare the intra-articular steroid administration with the extra-articular one; around the coracohumeral ligament in patients with adhesive capsulitis.

Method:

Ethics committee approval was obtained for the study. Patients who were diagnosed with adhesive capsulitis in the orthopedic outpatient clinic were included. Diagnosis was confimed by physical examination and Magnetic Resonance Imaging (MRI) findings. Patients with radiological finding of any tear in the rotator cuff or long head of biceps tendons were excluded. Only patients in the freezing or frozen stage of the disease were included. Patients who were previously treated with the diagnosis of adhesive caspulitis or who received any injections to the shoulder joint were not included in the study. Included patients were randomly divided into two groups according to age, sex, duration of complaint, concomitant diabetes mellitus (DM) disease and clinical stage of the disease. For randomization, stratified randomization was applied according to the information obtained from the outpatient clinic. While patients in group 1 received an anterior extra-articular steroid injection under USG guidance, patients in group 2 received posterior intra-articular steroid injection under USG guidance. A combination of 1 mL of triamcinolone acetonide (40 mg/mL) and 1 mL of prilocaine hydrochloride (2%) were injected to all patients. Patients were first evaluated before injection, than randomized to groups and prospectively followed up by an orthopaedic surgeon who was blinded to the groups. Evaluation was done for pain (visual analog scale score; VAS), functional status (American Shoulder and Elbow Surgeons score; ASES and Quick Disabilities of the Arm, Shoulder and Hand; Quick DASH), and active shoulder joint range of motion (ROM) angles at 1, 3, and 6 weeks after the injection. Means and standard deviations of were noted for each measurement period and each group. Improvements in each period between the groups and differences between the preinjection values and each follow-up period between the groups were analyzed using Ficher exact test, independent-samples t tests and Manova test. P < .05 was considered significant.

ELIGIBILITY:
Inclusion Criteria:

* must be between the ages of 18-75
* clinically and radiologically confirmed adhesive capsulitis

Exclusion Criteria:

* Patients with a tear in any of the rotator cuff tendons
* Patients who have had steroid injections in the shoulder region before
* patients who have been treated with the diagnosis of adhesive capsulitis (except for oral non-steroidal anti-inflammatory drug therapy)
* Patients with a previous history of trauma-fracture-dislocation in the shoulder region

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-05-24 (Estimated); Primary Completion 2024-11-24 (Estimated); Study Completion 2024-12-24 (Estimated)

PRIMARY OUTCOMES:
The Visual Analogue Scale(VAS) | The change from the baseline of the Visual Analog Scale (VAS) score of the shoulder pain in a period of 6 weeks Measurements will be taken at pre-medication, post-med 1.week, post-med 3.week, and post-med 6.week.
  The change of Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be'). Ask the patient to rate their current level of pain by placing a mark on the line.We noted the changes within this scoring system between the time framed which is stated below
external rotation of shoulder | The change from the baseline of external rotation of the shoulder in a period of 6 weeks Measurements will be taken at pre-medication, post-med 1.week, post-med 3.week, and post-med 6.week.
  The change of external rotation of the shoulder will be measured by the Orthopedic Resident by goniometer.
abduction of shoulder | The change in shoulder abduction from the baseline over a 6-week period Measurements will be taken at pre-medication, post-med 1.week, post-med 3.week, and post-med 6.week.
  The change of abduction of the shoulder will be measured by the Orthopedic Resident by goniometer.
flexion of shoulder | The change from the baseline of flexion of the shoulder in a period of 6 weeks Measurements will be taken at pre-medication, post-med 1.week, post-med 3.week, and post-med 6.week.
  The change of flexion of the shoulder will be measured by the Orthopedic Resident by a goniometer.
Internal rotation of the shoulder | The change from the baseline of internal rotation of the shoulder in a period of 6 weeks Measurements will be taken at pre-medication, post-med 1.week, post-med 3.week, and post-med 6.week.
  The change of Internal rotation of the shoulder will be measured by the Orthopedic Resident by Constant Shoulder Score

CONTACTS AND LOCATIONS:
Locations (1):
- Kartal Dr Lutfi Kirdar City Hospital, Istanbul, Kartal, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All the criteria specified and to be observed regarding the study will be transferred to the system in a timely manner and will be observed by the researchers outside the personal information of the patients.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: There will be no time limitations on data monitoring